CLINICAL TRIAL: NCT01809782
Title: Post-operative Cognitive Dysfunction (POCD) and Delirium in Patients Undergoing Two-stage Liver Operation - a Pilotstudy
Brief Title: Cognitive Outcome After Two-stage Liver-Operation
Acronym: 2-StaLi
Status: Terminated | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine, CCM and CVK, Charité - Universitätsmedizin Berlin, Germany, Charite University, Berlin, Germany
Other Study IDs: Two-stage liver
Record Dates: First submitted 2013-02-26; First posted 2013-03-13 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Delirium and Post-operative Cognitive Dysfunction (POCD)
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group:20 patients undergoing two stage liver-operation: Patients undergo two liver operations.First surgery: insitu-split for induction of proliferation in the remaining liver tissue; Second surgery: resection of the liver Tumor (4 cognitive measurements: Baseline, 7 days, 3 months and 1 year)
- Control group: 20 patients (ASA class II/III): Relatives from study personel or patients from outpatient clinics from Charité in Berlin and surrounding area (4 cognitive measurements: Baseline, 7 days, 3 months and 1 year)

SUMMARY:
Cognitive outcome (delirium and post-operative cognitive deficiency) in patients undergoing two-time liver resection.

ELIGIBILITY:
Study Group:

Inclusion Criteria:

* Patients undergoing a planned elective in situ split liver operation with following resection after approximately ten days with or without additional elective surgery in the same session at the University Hospital, Campus Virchow-Klinikum of the Charité - University Medicine Berlin
* Patients aged greater than or equal to 18 years
* Patients of both genders
* Offered patient information and written informed consent
* No participation in another clinical trial according to the German Drug Law (AMG) during the trial and one month before inclusion

Exclusion Criteria:

* Lacking willingness to save and hand out pseudonymised data within the clinical study
* Accommodation in an institution due to an official or judicial order
* Staff of Charite University hospital Berlin, Virchow Klinikum
* Illiteracy
* Unability of German language use
* Visual and acoustical impairment
* core on the mini mental state examination (MMSE) at screening of 23 or less
* American Society of Anaesthesiologists (ASA) Classification greater than IV
* Ascertained psychiatric disease
* Intake of psychotropic drugs (including sleeping pills and Benzodiazepine)
* Symptomatic bradycardia
* Symptomatic heart rhythm disorder (arrhythmia)
* Coronary heart disease Canadian Society of Anaesthesiologists criteria (CSC) stadium IV or the presentation of a coronary heart disease that needs intervention

Control Group:

Inclusion criteria:

•Male and female ASA II/III patients, aged ≥ 18 years

Exclusion Criteria:

* Mini-Mental-State-Examination ≤ 23 Points
* Neuropsychiatric morbidity, which limits the conduction of the neurocognitive testing
* Taking psychothropic drugs (including sleep-inducing drug and benzodiazepine) on a regular basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients undergoing two stage liver-operations
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2017-04-16 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
POCD | At postoperative day 7 after second liver operation
  Measured by Cambridge Neurophysiological Test Automated Battery (CANTAB); calculated in relation to a healthy control group without intervention
Delirium | At postoperative day 7 after second liver operation
  Measured by Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV)

SECONDARY OUTCOMES:
Delirium | At postoperative day 7 after second liver operation
  Measured by Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) and Confusion Assessment Method (CAM) and Intensive Care Delirium Screening Checklist (ICDSC) and Delirium Detection Scale (DDS) and Delirium Rating Scale (DRS) and The Nursing Delirium Screening Scale (NU-DESC)
Change of POCD | Change from pre-operative (Baseline) up to 365 days after surgery
  Measured by Cambridge Neurophysiological Test Automated Battery (CANTAB) calculated in relation to a healthy control group without intervention
Simplifies Acute Physiology Score (SAPS II) | At postoperative day 7 after second liver operation
  Simplifies Acute Physiology Score (SAPS II)
Length of post-operative hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Post-anaesthesia Discharge Scoring Stay (PADSS)
Length of post-operative intensive care unit stay | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Criteria of internal standard operating procedures (SOP)
Pain | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Measured by Numeric Rating Scale (NRS) or Verbal Rating Scale (VRS) or Visual Analogue Scale (VAS) or Behavioural Pain Scale (BPS)
The rate of post-operative organ dysfunctions and complications | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Cerebral-, cardiovascular-, cardiac- pulmonary-, gastrointestinal- and renal dysfunctions
Incidence of systemic inflammatory response syndrome (SIRS) and infection | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Centers for Disease Control (CDC) and American Thoracic Society (ATS) criteria
Change of 36-item short form health survey (SF-36) | Change from pre-operative (Baseline) up to 365 days after surgery
  36-item short form health survey (SF-36)
Mortality | after 90 days, after 182 days and after 365 days
  postoperative survival
Acute Physiological and Chronic Health Evaluation (Apache II) | At postoperative day 7 after second liver operation
  Acute Physiological and Chronic Health Evaluation (Apache II)
Sequental Organ Failure Assessment (SOFA) | At postoperative day 7 after second liver operation
  Sequental Organ Failure Assessment (SOFA)
TISS | At postoperative day 7 after second liver operation
  Therapeutic Interventions Scoring System (TISS)
RASS | At postoperative day 7 after second liver operation
  Richmonds Agitation Sedations Scale (RASS)
GCS | At postoperative day 7 after second liver operation
  Glasgow Coma Scale (GCS)
RIFLE criteria | At postoperative day 7 after second liver operation
  Risk Injury Failure Loss End Stage Kidney Disease (RIFLE = risk (R), injury (I), and failure (F), sustained loss (L) and end-stage kidney disease (E))
Change of EuroQoL instrument (EQ-5D) | Change from pre-operative (Baseline) up to 365 days after surgery
  EuroQoL instrument (EQ-5D)
Change of Barthel Index(for Activities of Daily Living, ADL) | Change from pre-operative (Baseline) up to 365 days after surgery
  Barthel Index (for Activities of Daily Living, ADL)
Change of Instrumentelle Aktivität im täglichen Leben (IATL) | Change from pre-operative (Baseline) up to 365 days after surgery
  Instrumentelle Aktivität im täglichen Leben (IATL)
Change of Geriatric Depression Scale (GDS) | Change from pre-operative (Baseline) up to 365 days after surgery
  Geriatric Depression Scale (GDS)
Change of Cornell Depression Scale (CDS) | Change from pre-operative (Baseline) up to 365 days after surgery
  Cornell Depression Scale (CDS)
Change of Hospital Anxiety and Depression Scale deutsche Version (HADS-D) | Change from pre-operative (Baseline) up to 365 days after surgery
  Hospital Anxiety and Depression Scale deutsche Version (HADS-D)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine Campus Charité Mitte and Campus Virchow-Klinikum, Berlin, Germany